CLINICAL TRIAL: NCT07250685
Title: Subthalamic Nucleus Versus Globus Pallidal Internus Deep Brain Stimulation for Parkinson Disease
Acronym: Superior PD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhang Jianguo (Other Government)
Responsible Party: Sponsor-Investigator, Zhang Jianguo, Deputy Director of the Neurosurgery Center,Director of the Functional Neurosurgery Ward,Director of the Neural Function Laboratory, Beijing Municipal Administration of Hospitals
Organization: Beijing Municipal Administration of Hospitals (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HX-A-2025009
Record Dates: First submitted 2025-11-14; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: PD - Parkinson's Disease
Keywords: Parkinson's disease(PD); Deep Brain Stimulation(DBS); Subthalamic Nucleus(STN); Globus Pallidus Internus(GPi)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: prospective, multicenter, superiority, double-blind, randomized crossover control.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First STN-DBS group (Experimental): Treatment involves deep brain electrode implantation with the STN target stimulation protocol.Stimulator activation time: To avoid the impact of local cerebral edema and microlesional effects after electrode implantation on clinical efficacy assessment, the STN target stimulator will be activated at the first follow-up visit.Postoperative medication: During the study period, patients are not prohibited from using drug therapy. Existing therapeutic drugs may be adjusted or new drugs for Parkinson's disease may be added.At the second follow-up visit, patients will receive the GPi target stimulation protocol.At the third follow-up visit, patients will receive the simultaneous STN + GPi stimulation protocol.At the final follow-up visit, the most clinically satisfactory stimulation protocol will be selected based on the patient's specific condition.Washout period: All patients will switch to GPi target therapy 90 days after receiving STN target stimulation.
  Interventions: Device: STN-DBS stimulation; Device: GPi-DBS stimulation; Device: STN&GPi-DBS stimulation
- First GPi-DBS group (Active Comparator): Treatment involves deep brain electrode implantation with the GPi target stimulation protocol.Stimulator activation time: To avoid the impact of local cerebral edema and microlesional effects after electrode implantation on clinical efficacy assessment, the GPi target stimulator will be activated at the first follow-up visit.Postoperative medication: During the study period, patients are not prohibited from using drug therapy. Existing therapeutic drugs may be adjusted or new drugs for Parkinson's disease may be added.At the second follow-up visit, patients will receive the STN target stimulation protocol.At the third follow-up visit, patients will receive the simultaneous STN + GPi stimulation protocol.At the final follow-up visit, the most clinically satisfactory stimulation protocol will be selected based on the patient's specific condition.Washout period: All patients will switch to STN target therapy 90 days after receiving GPi target stimulation.
  Interventions: Device: STN-DBS stimulation; Device: GPi-DBS stimulation; Device: STN&GPi-DBS stimulation

INTERVENTIONS:
Device: STN-DBS stimulation — The devices for this study are provided by Boston Scientific International Medical Trading (Shanghai) Co., Ltd.The system consists of two components: electrodes and an implanted stimulator.Participants will be implanted with an 8-contact directional electrode (Model: DB-2202-45).The stimulator is a rechargeable model (Model: DB-1232).
  Participants will receive the STN target stimulation protocol for a 3-month treatment period.
Device: GPi-DBS stimulation — The devices for this study are provided by Boston Scientific International Medical Trading (Shanghai) Co., Ltd.The system consists of two components: electrodes and an implanted stimulator.Participants will be implanted with an 8-contact directional electrode (Model: DB-2202-45).The stimulator is a rechargeable model (Model: DB-1232).
  Participants will receive the GPi target stimulation protocol for a 3-month treatment period.
Device: STN&GPi-DBS stimulation — The devices for this study are provided by Boston Scientific International Medical Trading (Shanghai) Co., Ltd.The system consists of two components: electrodes and an implanted stimulator.Participants will be implanted with an 8-contact directional electrode (Model: DB-2202-45).The stimulator is a rechargeable model (Model: DB-1232).
  After participants receive 3 months of STN target monotherapy and 3 months of GPi target monotherapy sequentially, they will be administered the combined STN + GPi target stimulation protocol. Prior to the initiation of simultaneous STN + GPi stimulation, participants are required to turn off the stimulator for 4 hours to eliminate the residual effects of the previous target stimulation.

SUMMARY:
The primary objective of this prospective, multicenter, double-blind, randomized, crossover clinical trial is to evaluate whether Subthalamic Nucleus-Deep Brain Stimulation (STN-DBS) is more effective than Globus Pallidus Internus-Deep Brain Stimulation (GPi-DBS) in improving motor symptoms of patients with Parkinson's disease at 90 days post-treatment.

DETAILED DESCRIPTION:
The primary objective of this prospective, multicenter, double-blind, randomized crossover controlled clinical trial is to evaluate whether STN-DBS provides superior efficacy over GPi-DBS in improving motor symptoms of Parkinson's disease patients at 90 days post-treatment.

Randomization of this study is generated by a centralized Contract Research Organization (CRO). At the second follow-up visit, patients will be assigned according to the randomization code list in the system, with each patient first receiving either STN-DBS or GPi-DBS. The randomization ratio between the two groups is 1:1. At the third follow-up visit, each group will then receive stimulation at the other target.

Assessments of motor function, cognitive level, anxiety and depression status, and quality of life will be conducted preoperatively. The device will be activated 30 days postoperatively. Target adjustments, along with assessments of motor function, cognitive level, anxiety and depression status, quality of life, and adverse events, will be performed at 120, 210, and 300 days postoperatively.

The grouping information will only be known to the operating surgeons and programming physicians, while other investigators, assessing physicians, and patients will remain blinded. This study will be completed within 24 months, enrolling 86 patients from 7 centers in China, with 43 patients in each group. The Data Safety Monitoring Board (DSMB) will conduct regular monitoring to ensure the safe conduct of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age at the time of enrollment: 22-75 years.
2. Diagnosis of bilateral idiopathic PD with the presence of at least 2 of the following: resting tremor, rigidity, or bradykinesia
3. Duration of idiopathic PD: ≥ 5 years.
4. Severity of PD in the meds off condition: Hoehn-Yahr stages 2.5~ 4.0.
5. Despite optimal medication treatment, there are still persistent symptoms or drug side effects of disabling Parkinson's
6. Must have tried a form of carbidopa/levodopa and/or one of the dopamine agonists as part of medication therapy.
7. Anti-parkinsonian medications must improve PD symptoms by ≥33%, as measured by UPDRS-III score.
8. UPDRS-III score of ≥ 30 in the meds off condition.
9. The MMSE assessment was higher than the demarcation score of the corresponding educational level, and the cognitive function was normal.
10. HAMD score≤24.
11. No change in antidepressant medications utilized for treatment of depression for at least 8 weeks prior to informed consent.
12. Stable on anti-parkinsonian medication for 28 days prior to informed consent.
13. Could tolerate bilateral STN DBS and bilateral GPi DBS.
14. Be willing and able to comply with all visits and study related procedures (e.g., using the remote control, charging system and completing the PD Diary
15. Able to understand the study requirements and the treatment procedures and provides written informed consent before any studyspecific tests or procedures are performed.

Exclusion Criteria:

1. Any intracranial abnormalities or medical conditions that Lead to the prohibition of DBS surgery.
2. Have any significant psychiatric condition likely to compromise the subject's ability to comply with requirements of the study protocol (e.g. bipolar, schizophrenia, mood disorder with psychotic features, cluster B personality disorders).
3. HAMD score>24.
4. Any current drug or alcohol abuse, per DSM-IV criteria
5. Any history of recurrent or unprovoked seizures.
6. Any history of hemorrhagic stroke.
7. Any previous treatment for movement disorders involving intracranial surgery or device implantation.
8. Any other active implanted devices including neurostimulators (e.g., cochlear implant, pacemaker) and /or drug delivery pumps, whether turned on or off. Passive implants (e.g., knee prostheses) would be allowed provided that they do not interfere with the functioning of the DBS system
9. Any previous thalamotomy, pallidotomy or subjects who have undergone a DBS procedure.
10. Any previously implanted Vagus Nerve Stimulation (VNS) patients.
11. Any previous brain surgery that would interfere with the placement of the leads or the functioning of the device.
12. A condition requiring or likely to require the use of Magnetic Resonance Imaging (MRI), diathermy or electroconvulsive therapy (ECT)
13. Likely to require the use of monopolar cau Likely to require the use of monopolar cautery, radiofrequency (RF) procedures, external defibrillation, lithotripsy, radiation therapy or transcranial stimulation.tery, radiofrequency (RF) procedures, external defibrillation, lithotripsy, radiation therapy or transcranial stimulation.
14. Currently on any anticoagulant medications that cannot be discontinued during perioperative period.
15. Currently exhibiting secondary Parkinsonism due to prescribed medications.
16. Have any significant medical condition that is likely to interfere with study procedures or likely to confound evaluation of study endpoints.
17. Any terminal illness with life expectancy of < 1 year.
18. Any unresolved infection, a coagulopathy or significant cardiac or other medical risk factor for surgery
19. Current or future risk of being immunocompromised that might significantly increase risk of infection.
20. Participation in any other clinical trial (e.g. drug, device, or biologics) concurrently or within the preceding 30 days. Participation in any other study will be allowed per investigator/sponsor discretion only.
21. A female who is breastfeeding or of child-bearing potential with a positive urine pregnancy test or not using adequate contraception.
22. Preoperative DBS plan failed to implant STN and GPi. nuclei.(Usually limited by individual anatomical differences)
23. Preoperative CT scan of the head revealed calcification of the GPI.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-11-24 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale Part III (UPDRS III) score | Before surgery and 90 days (±7 days) after surgery
  The differences in UPDRS III scores obtained under the stimulation state at 90 days (±7 days) after surgery, compared with the preoperative scores, in patients with Parkinson's disease who received Subthalamic Nucleus-Deep Brain Stimulation (STN-DBS) or Globus Pallidus Internus-Deep Brain Stimulation (GPi-DBS) treatment.
  Doctors conducted double-blind evaluations based on this scoring scale. The Unified Parkinson's Disease Rating Scale Part III (UPDRS III) has a scoring range of 0 to 108 points, with higher scores indicating more severe motor symptoms in patients with Parkinson's disease.

SECONDARY OUTCOMES:
Freezing of Gait Questionnaire (FOG-Q) score | Before surgery and 90 days (±7 days) after surgery
  Description: The differences in FOG-Q scores obtained under the stimulation state at 90 days (±7 days) after surgery, compared with the preoperative scores, in patients with Parkinson's disease who received Subthalamic Nucleus-Deep Brain Stimulation (STN-DBS) or Globus Pallidus Internus-Deep Brain Stimulation (GPi-DBS) treatment. Doctors conducted evaluations based on this scoring scale. The Freezing of Gait Questionnaire (FOG-Q) has a scoring range of 0 to 24 points, with higher scores indicating more severe freezing of gait symptoms.
Berg Balance Scale (BBS) score | Before surgery and 90 days (±7 days) after surgery
  Description: The differences in BBS scores obtained under the stimulation state at 90 days (±7 days) after surgery, compared with the preoperative scores, in patients with Parkinson's disease who received STN-DBS or GPi-DBS treatment. Doctors conducted evaluations based on this scoring scale. The Berg Balance Scale (BBS) has a scoring range of 0 to 56 points, with higher scores indicating better balance function.
Unified Dyskinesia Rating Scale (UDysRS) score | Before surgery and 90 days (±7 days) after surgery
  The differences in UDysRS scores obtained under the stimulation state at 90 days (±7 days) after surgery, compared with the preoperative scores, in patients with Parkinson's disease who received STN-DBS or GPi-DBS treatment. Doctors conducted evaluations based on this scoring scale. The Unified Dyskinesia Rating Scale (UDysRS) has a scoring range of 0 to 104 points, with higher scores indicating more severe dyskinesia symptoms.
Mini-Mental State Examination (MMSE) score | Before surgery and 90 days (±7 days) after surgery
  The differences in MMSE scores obtained under the stimulation state at 90 days (±7 days) after surgery, compared with the preoperative scores, in patients with Parkinson's disease who received STN-DBS or GPi-DBS treatment. Doctors conducted evaluations based on this scoring scale. The Mini-Mental State Examination (MMSE) has a scoring range of 0 to 30 points, with higher scores indicating better cognitive function.
Montreal Cognitive Assessment (MoCA) score | Before surgery and 90 days (±7 days) after surgery
  The differences in MoCA scores obtained under the stimulation state at 90 days (±7 days) after surgery, compared with the preoperative scores, in patients with Parkinson's disease who received STN-DBS or GPi-DBS treatment. Doctors conducted evaluations based on this scoring scale. The Montreal Cognitive Assessment (MoCA) has a scoring range of 0 to 30 points, with higher scores indicating better cognitive function (a score ≥26 is considered normal).
Hamilton Anxiety Rating Scale (HAMA) score | Before surgery and 90 days (±7 days) after surgery
  The differences in HAMA scores obtained under the stimulation state at 90 days (±7 days) after surgery, compared with the preoperative scores, in patients with Parkinson's disease who received STN-DBS or GPi-DBS treatment. Doctors conducted evaluations based on this scoring scale. The Hamilton Anxiety Rating Scale (HAMA) has a scoring range of 0 to 56 points, with higher scores indicating more severe anxiety symptoms.
Hamilton Rating Scale for Depression (HRSD) score | Before surgery and 90 days (±7 days) after surgery
  The differences in HRSD scores obtained under the stimulation state at 90 days (±7 days) after surgery, compared with the preoperative scores, in patients with Parkinson's disease who received STN-DBS or GPi-DBS treatment. Doctors conducted evaluations based on this scoring scale. The Hamilton Rating Scale for Depression (HRSD) has a scoring range of 0 to 52 points, with higher scores indicating more severe depressive symptoms.
Parkinson's Disease Questionnaire-39 (PDQ-39) score | Before surgery and 90 days (±7 days) after surgery
  The differences in PDQ-39 scores obtained under the stimulation state at 90 days (±7 days) after surgery, compared with the preoperative scores, in patients with Parkinson's disease who received STN-DBS or GPi-DBS treatment. Patients completed the questionnaire for evaluation. The Parkinson's Disease Questionnaire-39 (PDQ-39) is scored as a summary index (0-156), with higher scores indicating poorer quality of life.
Programming parameters | 90 days (±7 days) after surgery
  The differences in programming parameters (including Total Electrical Energy Delivered [TEED], contact, current, pulse width, and frequency) at 90 days (±7 days) after surgery between Parkinson's disease patients who received STN-DBS or GPi-DBS treatment.
Differences in programming parameters and medication under combined stimulation | Baseline and 90 days (±7 days) after surgery
  The differences in programming parameters (including UPDRS III score, TEED, contact, voltage, pulse width, frequency) and medication (Levodopa Equivalent Daily Dose [LEDD]) at 90 days (±7 days) after surgery, compared with baseline, in Parkinson's disease patients receiving simultaneous STN-DBS and GPi-DBS treatment.
Patient preference for stimulation targets | 90 days (±7 days) after surgery
  Patient preference for activated stimulation targets under three conditions: STN-DBS alone, GPi-DBS alone, and simultaneous STN-DBS and GPi-DBS.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Beijing Tiantan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Nanjing Brain Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sidiropoulos C, LeWitt PA, Odekerken VJ, Schuurman PR, de Bie RM. GPi vs STN deep brain stimulation for Parkinson disease: Three-year follow-up. Neurology. 2016 Aug 16;87(7):745-6. doi: 10.1212/WNL.0000000000003027. No abstract available. PMID 27527541
- [Result] Xu H, Zheng F, Krischek B, Ding W, Xiong C, Wang X, Niu C. Subthalamic nucleus and globus pallidus internus stimulation for the treatment of Parkinson's disease: A systematic review. J Int Med Res. 2017 Oct;45(5):1602-1612. doi: 10.1177/0300060517708102. Epub 2017 Jul 12. PMID 28701061
- [Result] Dulski J, Schinwelski M, Konkel A, Grabowski K, Libionka W, Waz P, Sitek EJ, Slawek J. The impact of subthalamic deep brain stimulation on sleep and other non-motor symptoms in Parkinson's disease. Parkinsonism Relat Disord. 2019 Jul;64:138-144. doi: 10.1016/j.parkreldis.2019.04.001. Epub 2019 Apr 5. PMID 30975618
- [Result] Ramirez-Zamora A, Ostrem JL. Globus Pallidus Interna or Subthalamic Nucleus Deep Brain Stimulation for Parkinson Disease: A Review. JAMA Neurol. 2018 Mar 1;75(3):367-372. doi: 10.1001/jamaneurol.2017.4321. PMID 29356826
- [Result] Okun MS. Deep-brain stimulation--entering the era of human neural-network modulation. N Engl J Med. 2014 Oct 9;371(15):1369-73. doi: 10.1056/NEJMp1408779. Epub 2014 Sep 8. No abstract available. PMID 25197963
- [Result] Chen J, Liu JL, Chen X, Qian H, Xian WB, Zhou HY, Liu YM, Ye XF, Zheng YF, Zhang SL, Chen L, Li JR, Liu ZL, Pei Z. [Significant improvement of motor symptoms by deep brain stimulation of bilateral subthalamic nucleus in patients with moderate or advanced Parkinson's disease]. Zhonghua Yi Xue Za Zhi. 2011 Feb 1;91(5):291-5. Chinese. PMID 21419000
- [Result] Nova IC, Perracini MR, Ferraz HB. Levodopa effect upon functional balance of Parkinson's disease patients. Parkinsonism Relat Disord. 2004 Oct;10(7):411-5. doi: 10.1016/j.parkreldis.2004.04.004. PMID 15465397
- [Result] Bejjani BP, Gervais D, Arnulf I, Papadopoulos S, Demeret S, Bonnet AM, Cornu P, Damier P, Agid Y. Axial parkinsonian symptoms can be improved: the role of levodopa and bilateral subthalamic stimulation. J Neurol Neurosurg Psychiatry. 2000 May;68(5):595-600. doi: 10.1136/jnnp.68.5.595. PMID 10766889
- [Result] Ma CL, Su L, Xie JJ, Long JX, Wu P, Gu L. The prevalence and incidence of Parkinson's disease in China: a systematic review and meta-analysis. J Neural Transm (Vienna). 2014 Feb;121(2):123-34. doi: 10.1007/s00702-013-1092-z. Epub 2013 Sep 22. PMID 24057652